CLINICAL TRIAL: NCT07010744
Title: Effect of Triple Versus Quadruple Therapy for Treating Helicobacter Pylori Infection -an Open Label Randomized Controlled Trial
Brief Title: Effect of Triple Versus Quadruple Therapy for Treating Helicobacter Pylori Infection
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Akil Al Islam (Other)
Responsible Party: Sponsor-Investigator, Akil Al Islam, Principal Investigator, Dhaka Medical College
Organization: Dhaka Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-DMC/2025/39
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple drug Therapy (Experimental): Triple drug therapy includes Amoxicillin , clarithromycin and esomeprazole
  Interventions: Drug: Triple drug regimen
- Quadruple therapy (Experimental): Bismuth Metronidazole Tetracycline Esomeprazole
  Interventions: Drug: Quadruple therapy

INTERVENTIONS:
Drug: Triple drug regimen — Amoxicillin 1000mg at 12 hourly for 14 days Clarithromycin 500mg at 12 hourly for 14 days Esomeprazole 20 mg at 12 hourly for 14 days
  Arms: Triple drug Therapy
Drug: Quadruple therapy — Bismuth subcitrate 120 mg at 6 hourly 14 days Metronidazole 500mg at 8 hourly 14 days Tetracycline 500mg at 6 hourly 14 days Esomeprazole 20 mg 12 hourly for 14 days
  Arms: Quadruple therapy

SUMMARY:
The Goal of this this clinical trial is to assess and compare the eradication rate of triple and quadruple therapy during treating helicobacter pylori infection among patients presented with dyspepsia. It will also assess the patient reported adverse events among two groups.

H pylori infection will be confirmed by CLO (RUT) test and stool antigen test both.

Standard triple therapy will be based on Esomeprazole 20 mg BD, Clarithromycin 500mg BD and Amoxicillin 1gm BD. Bismuth Quadruple therapy consists of Bismuth subsalicylate 300mg QDS, Tetracycline 500mg QDS and Metronidazole 400mg TDS. Patient will be confirmed H pylori eradication 4 weeks after completion of treatment by Stool antigen test only.

DETAILED DESCRIPTION:
This Randomized Controlled Trial study aims to compare the eradication rates of Helicobacter pylori infection between quadruple therapy and triple therapy in dyspeptic patients at Dhaka Medical College & Hospital.

Sixty-Six participants, selected through purposive sampling, will be randomly allocated into two groups: 33 patients in Group A (receiving Triple therapy) and 33 in Group B (receiving Quadruple therapy). After pre-procedural preparation, a CLO test will be conducted during endoscopy and a stool antigen test to detect H. pylori. Participants will undergo treatment for 14 days, followed by follow-up testing 4 weeks later to evaluate eradication. Ethical approval will be obtained, and confidentiality will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* All dyspeptic patients aged ≥18 years.
* Patients who will provide informed written consent and agree to follow-up at 4 weeks post-treatment.

Exclusion Criteria:

* Patients who have received prior H. pylori eradication therapy.
* Ingestion of antibiotics or proton pump inhibitor within the prior 4 weeks. Patient who will test negative either of CLO or Stool Antigen Test or both
* Patients with known allergies or intolerance to any of the study medications.
* Patients with alarm symptoms (e.g., unexplained weight loss, persistent vomiting, dysphagia).
* Patients with a history of gastric surgery.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To compare the eradication rate of Helicobacter pylori infection between quadruple therapy and triple therapy among dyspeptic patients | 1 month

SECONDARY OUTCOMES:
1. To determine the eradication rate of H. pylori in patients receiving triple drug therapy. 2. To determine the eradication rate of H. pylori in patients receiving quadruple therapy. 3. Assess and quantify patient reported adverse events in both groups | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Akil Al Islam, MBBS,MRCP, Principal Investigator — Dhaka Medical College
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
I shall decide it later